CLINICAL TRIAL: NCT02313701
Title: Effect of Standardized Consent for Urogynecological Procedures on Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Roger Lefevre, Instructor in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2014P000273
Record Dates: First submitted 2014-11-10; First posted 2014-12-10 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Vaginal hysterectomy counseling (No Intervention): Standard verbal counseling to consent for vaginal hysterectomy in terms of what the procedures involves, other treatment options, risks, benefits, and what to expect in the pre-op and post-op periods. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
- Vaginal hysterectomy visual aid (Experimental): In addition to standard verbal counseling, intervention will include a standardized visual presentation for vaginal hysterectomy. Time spent viewing the visual presentation will be recorded to assess for the efficiency of this quality improvement intervention. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
  Interventions: Other: Standardized visual presentation
- Robotic sacrocolpopexy counseling (No Intervention): Standard verbal counseling to consent for robotic sacrocolpopexy in terms of what the procedures involves, other treatment options, risks, benefits, and what to expect in the pre-op and post-op periods. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
- Robotic sacrocolpopexy visual aid (Experimental): In addition to standard verbal counseling, intervention will include a standardized visual presentation for robotic sacrocolpopexy. Time spent viewing the visual presentation will be recorded to assess for the efficiency of this quality improvement intervention. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
  Interventions: Other: Standardized visual presentation
- Sub-urethral sling counseling (No Intervention): Standard verbal counseling to consent for sub-urethral sling in terms of what the procedures involves, other treatment options, risks, benefits, and what to expect in the pre-op and post-op periods. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
- Sub-urethral sling visual aid (Experimental): In addition to standard verbal counseling, intervention will include a standardized visual presentation for sub-urethral sling. Time spent viewing the visual presentation will be recorded to assess for the efficiency of this quality improvement intervention. At the end of the clinic visit, participants will receive a survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.
  Interventions: Other: Standardized visual presentation

INTERVENTIONS:
Other: Standardized visual presentation — Visual presentations will address what type of procedure they will undergo, the risks and benefits of the procedure (i.e. injury to nearby organs, risks of infection and bleeding, risk of re-operation), alternative treatments to the procedure, what to expect during the pre-operative period, and what to expect in the post-operative period (i.e. urinary catheter, constipation, pain management, hospital stay).
  Arms: Robotic sacrocolpopexy visual aid; Sub-urethral sling visual aid; Vaginal hysterectomy visual aid

SUMMARY:
The investigators aim is to augment the current process for surgical consent for patients undergoing urogynecological procedures by incorporating visual media. We propose that visual media will be an effective and efficient addition to the standard of care in urogynecological consents and will improve patient understanding and satisfaction. Our randomized controlled trial will investigate the effect of standardizing the consent for three urogynecologic procedures (vaginal hysterectomy, robotic sacrocolpopexy, and sub-urethral sling) using visual media, on patients' understanding of, and satisfaction with, their procedure. Our primary outcome will be patient's knowledge score at the end of the pre-operative clinic visit, and secondary outcomes include patients' satisfaction, subjective understanding of their procedure, immediate pre-operative and post-operative knowledge, and number of post-operative encounters. Participants will be followed up to their post-operative clinic visit.

DETAILED DESCRIPTION:
Background

The current standard of care for consenting patients undergoing urogynecological procedures involves counseling patients on the procedures, other treatment options, risks, benefits, and pre-op and post-op periods. This counseling is routinely done verbally and may not be consistently standardized across patients. Pre-operatively, patients may undergo testing and post-operatively, patients may be admitted to the hospital and/or discharged with a urinary catheter following a voiding trial. Patients may also experience pain and constipation post-operatively at the hospital or at home and in the long term may experience recurrence of their symptoms and require reoperation.

The existing literature cites many examples of quality improvement initiatives and studies focused on improving the surgical consent process, patients' understanding and satisfaction. Several systematic reviews include prospective and randomized controlled trials using various patient counseling interventions including videos, computer programs, electronic presentation, websites, powerpoint, and written information have found improved patient comprehension and knowledge but did not consistently affect satisfaction (Farrell et al. Patient Education and Counseling. 2012;94:20-32. Nehme et al. Surg Innov. 2013;20(1):13-23. Schenker et al. Med Decis Making. 2011;31:151-173.). Most trials reported outcomes including overall satisfaction, knowledge score, perceived understanding (Hoppe et al. J Shoulder Elbow Surg. 2014;23:e134-e139. Johannes et al. Ann Surg Oncol. 2013;20:15-23. Bollschweiler et al. Ann Surg. 2008;258:205-211.). However, there has not been any such prospective randomized controlled trial for improving the consent process using media aid for urogynecological procedures. A related prospective study reported patients' understanding of sacrocolpopexy without any intervention and found deficiencies with mean knowledge score of less than 70 out of 100 (Adams et al. Female Pelvic Med Reconstr Surg. 2012;18(6):352-356.).

In our study, we hope to incorporate and assess the effectiveness of standardized visual presentation in addition to the standard of care. We hope to use the results of our study to inform our clinical practice and improve our patients' understanding and satisfaction.

Design and Overview

Our randomized controlled trial will investigate the effect of standardizing the consent for three urogynecologic procedures (vaginal hysterectomy, robotic sacrocolpopexy, and sub-urethral sling) using visual media, on patients' understanding of, and satisfaction with, their procedure.

Eligible patients will be recruited by a member of the research team at their pre-operative clinic visits. Participants who decline to enroll will not have access to the additional materials, but will receive the same standard level of care as the enrolled participants.

Currently, the standard of care for consenting patients for these three procedures involves verbally counseling patients on what the procedures involves, other treatment options, risks, benefits, and what to expect in the pre-op and post-op periods. In this study, for each of the three surgical procedures, we will use a computer-generated scheme to allocate participants in a 1:1 ratio using block randomization. Participants will be randomized to one of two study arms:

1. Participants will receive the standard counseling described above
2. Participants will receive the same counseling as described above and will then review a standardized visual presentation for the procedure they will undergo.

Each participant will be first provided the standard of care that they would have received at a pre-operative clinic visit. Then, participants in the intervention arm will view a visual presentation that will address what type of procedure they will undergo, the risks and benefits of the procedure (i.e. injury to nearby organs, risks of infection and bleeding, risk of re-operation), alternative treatments to the procedure, what to expect during the pre-operative period, and what to expect in the post-operative period (i.e. urinary catheter, constipation, pain management, hospital stay). Time spent viewing the visual presentation will be recorded to assess for the efficiency of this quality improvement intervention. At the end of the clinic visit, all participating patients will receive the same survey to evaluate their understanding of their procedure, pre-operative and post-operative expectations, and satisfaction with their experience. A similar survey will be repeated before their surgery and at their post-operative clinic visit at approximately 1-2 weeks following the surgery.

Outcome Ascertainment

Our primary outcome will be patient's knowledge score at the end of the pre-operative clinic visit, and secondary outcomes include patients' satisfaction, subjective understanding of their procedure, immediate pre-operative and post-operative knowledge, and number of post-operative encounters. Participants will be followed up to their post-operative clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing vaginal hysterectomy, robotic sacrocolpopexy, or sub-urethral sling
* English speaking
* Written, informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Patient knowledge score | Within 8 hours of pre-operative clinic visit, which can be up to 10 weeks from time of enrollment
  At the end of the clinic visit, all participating patients will receive a survey to evaluate their objective understanding of their procedures, pre-operative and post-operative expectations.

SECONDARY OUTCOMES:
Patient satisfaction | Within 8 hours of pre-operative clinic visit, which can be up to 10 weeks from time of enrollment
  At the end of the clinic visit, all participating patients will receive a survey to evaluate their satisfaction with their experience.
Patient subjective understanding of their procedures | Within 8 hours of pre-operative clinic visit, which can be up to 10 weeks from time of enrollment
  At the end of the clinic visit, all participating patients will receive a survey to evaluate their subjective understanding of their procedures, pre-operative and post-operative expectations.
Immediate pre-operative knowledge score | Within 24 hours prior to time of surgery
  Before their surgeries, all participating patients will receive a survey to evaluate their understanding of their procedures, pre-operative and post-operative expectations.
Post-operative knowledge score | Within 8 hours after routine post-operative visit, which is on average within 2 weeks after the time of surgery
  At the end of the clinic visit, all participating patients will receive a survey to evaluate their understanding of their procedures, pre-operative and post-operative expectations.
Number of post-operative encounters | Followed until scheduled routine post-operative visit, average of 2 weeks after time of surgery
  Number of post-operative encounters including telephone encounters and non-routine visits between the time of surgery and the routine post-operative clinic visit, which is scheduled when surgery is booked, will be recorded from patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Lefevre, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams SR, Hacker MR, Merport Modest A, Rosenblatt PL, Elkadry EA. Informed consent for sacrocolpopexy: is counseling effective in achieving patient comprehension? Female Pelvic Med Reconstr Surg. 2012 Nov-Dec;18(6):352-6. doi: 10.1097/SPV.0b013e31827816c5. PMID 23143430
- [Background] Nehme J, El-Khani U, Chow A, Hakky S, Ahmed AR, Purkayastha S. The use of multimedia consent programs for surgical procedures: a systematic review. Surg Innov. 2013 Feb;20(1):13-23. doi: 10.1177/1553350612446352. Epub 2012 May 14. PMID 22589017
- [Background] Schenker Y, Fernandez A, Sudore R, Schillinger D. Interventions to improve patient comprehension in informed consent for medical and surgical procedures: a systematic review. Med Decis Making. 2011 Jan-Feb;31(1):151-73. doi: 10.1177/0272989X10364247. Epub 2010 Mar 31. PMID 20357225
- [Derived] Wang R, Haviland MJ, Hacker MR, Lefevre R. Effect of Visual Aids During Surgical Consents on Patient Understanding and Satisfaction. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):746-750. doi: 10.1097/SPV.0000000000000703. PMID 31135580